CLINICAL TRIAL: NCT05418608
Title: Novel in Vivo Synaptic Imaging in Experienced Meditators
Acronym: app311_med
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000030601; 1R21AT011575-01 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Behavior, Health
Keywords: Meditation; Experienced meditators
MeSH Terms: conditions — Health Behavior | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aim 1 (Experimental): A PET study of the novel SV2A imaging tracer [11C]UCB-J in participants, to characterize the distribution of [11C]UCB-J in cortical and subcortical areas in experienced meditators compared to non-meditating controls. Subjects will undergo one PET scan with [11C]UCB-J and one MRI scan for anatomical identification of brain regions.
  Interventions: Drug: Radiotracer

INTERVENTIONS:
Drug: Radiotracer — A novel SV2A imaging tracer which is used in conjunction with positron emission tomography scans.
  Other Names: [11C]APP311; [11C]UCB-J

SUMMARY:
To utilize positron emission tomography (PET) imaging to characterize the distribution of (aka [11C]APP311at the Yale PET Center) in cortical and subcortical areas in experienced meditators compared to non-meditating controls.

DETAILED DESCRIPTION:
The investigators will conduct a PET study of the novel SV2A imaging tracer [11C]UCB-J in participants, to characterize the distribution of [11C]UCB-J in cortical and subcortical areas in experienced meditators compared to non-meditating controls. A total of up to 20 subjects will complete the study. Subjects will undergo one PET scan with [11C]UCB-J. Each subject will also undergo one MRI scan for anatomical identification of brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Age 28-70 years
* Voluntary, written, informed consent
* Physically healthy by medical history, physical, ECG and laboratory examinations
* At least 10 years and 5,000 hours of regular meditation practice
* For females, non-lactating, no longer of child-bearing potential or agree to practice effective contraception during the study, as well as a negative serum pregnancy (β-HCG) test at screening, and negative urine pregnancy on PET scanning days.

Exclusion Criteria:

* A history of significant psychiatric, medical (e.g., cardiovascular, renal) or neurological (e.g., cerebrovascular, seizure, traumatic brain injury) illness that is unstable and/or might affect the study objectives.
* Current or history of substance dependence (e.g., alcohol, nicotine, opiates, sedative hypnotics, etc.)
* Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
* Subjects with current, past or anticipated exposure to radiation in the work place within one year of proposed research PET scans that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits.
* Medical contraindications to participation in a magnetic resonance imaging procedure (e.g., ferromagnetic implants/foreign bodies, claustrophobia, cardiac pacemaker, prosthetic valve, otologic implant, etc.)
* History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).
* Medications that effect SV2A binding (e.g., levetiracetam).

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Analyzing positron emission tomography images in conjunction with magnetic resonance data | Up to two years
  Imaging data will be analyzed by using kinetic modeling approaches; these are used to quantitate total tracer binding, volume of distribution, and binding potential, specifically voxel-by-voxel compartment model fitting with the arterial input function. Positron emission tomography (PET) images will be registered to the subject's T1-weighted magnetic resonance (MR) images, and then registered to an magnetic resonance template. Gray matter regions of interest are determined by combining a predefined set of regions, defined on the template (Anatomical Automatic Labeling (AAL) for SPM2) with the gray matter segmentation mask (FAST algorithm in FSL). This process will permit direct, automatic determination of outcome values. Partial volume correction will also be applied to account for atrophy. Magnetic resonance (MR) image analyses will be done by standardized methods.

SECONDARY OUTCOMES:
Evaluating the correlation between data collected from meditation questionnaires and synaptic vesicle glycoprotein 2 (SV2A) binding | Up to two years
  Meditation assessments collected from participants, containing mindfulness and attention measures, will be correlated with synaptic vesicle glycoprotein 2 (SV2A) binding data, collected during a positron emission tomography scan.

CONTACTS AND LOCATIONS:
Overall Officials: David Matuskey, MD, Principal Investigator — Yale University
Locations (1):
- Yale University PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nabulsi NB, Mercier J, Holden D, Carre S, Najafzadeh S, Vandergeten MC, Lin SF, Deo A, Price N, Wood M, Lara-Jaime T, Montel F, Laruelle M, Carson RE, Hannestad J, Huang Y. Synthesis and Preclinical Evaluation of 11C-UCB-J as a PET Tracer for Imaging the Synaptic Vesicle Glycoprotein 2A in the Brain. J Nucl Med. 2016 May;57(5):777-84. doi: 10.2967/jnumed.115.168179. Epub 2016 Feb 4. PMID 26848175
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Ospina MB, Bond K, Karkhaneh M, Tjosvold L, Vandermeer B, Liang Y, Bialy L, Hooton N, Buscemi N, Dryden DM, Klassen TP. Meditation practices for health: state of the research. Evid Rep Technol Assess (Full Rep). 2007 Jun;(155):1-263. PMID 17764203
- [Background] Marchand WR. Neural mechanisms of mindfulness and meditation: Evidence from neuroimaging studies. World J Radiol. 2014 Jul 28;6(7):471-9. doi: 10.4329/wjr.v6.i7.471. PMID 25071887
- [Background] Ivanovski B, Malhi GS. The psychological and neurophysiological concomitants of mindfulness forms of meditation. Acta Neuropsychiatr. 2007 Apr;19(2):76-91. doi: 10.1111/j.1601-5215.2007.00175.x. PMID 26952819
- [Background] Marchand WR. Mindfulness-based stress reduction, mindfulness-based cognitive therapy, and Zen meditation for depression, anxiety, pain, and psychological distress. J Psychiatr Pract. 2012 Jul;18(4):233-52. doi: 10.1097/01.pra.0000416014.53215.86. PMID 22805898
- [Background] Afonso RF, Kraft I, Aratanha MA, Kozasa EH. Neural correlates of meditation: a review of structural and functional MRI studies. Front Biosci (Schol Ed). 2020 Mar 1;12(1):92-115. doi: 10.2741/S542. PMID 32114450
- [Background] Brewer JA, Worhunsky PD, Gray JR, Tang YY, Weber J, Kober H. Meditation experience is associated with differences in default mode network activity and connectivity. Proc Natl Acad Sci U S A. 2011 Dec 13;108(50):20254-9. doi: 10.1073/pnas.1112029108. Epub 2011 Nov 23. PMID 22114193
- [Background] Raichle ME. The brain's default mode network. Annu Rev Neurosci. 2015 Jul 8;38:433-47. doi: 10.1146/annurev-neuro-071013-014030. Epub 2015 May 4. PMID 25938726
- [Background] Northoff G, Heinzel A, de Greck M, Bermpohl F, Dobrowolny H, Panksepp J. Self-referential processing in our brain--a meta-analysis of imaging studies on the self. Neuroimage. 2006 May 15;31(1):440-57. doi: 10.1016/j.neuroimage.2005.12.002. Epub 2006 Feb 7. PMID 16466680
- [Background] Fox KC, Nijeboer S, Dixon ML, Floman JL, Ellamil M, Rumak SP, Sedlmeier P, Christoff K. Is meditation associated with altered brain structure? A systematic review and meta-analysis of morphometric neuroimaging in meditation practitioners. Neurosci Biobehav Rev. 2014 Jun;43:48-73. doi: 10.1016/j.neubiorev.2014.03.016. Epub 2014 Apr 3. PMID 24705269
- [Background] Van Dam NT, van Vugt MK, Vago DR, Schmalzl L, Saron CD, Olendzki A, Meissner T, Lazar SW, Kerr CE, Gorchov J, Fox KCR, Field BA, Britton WB, Brefczynski-Lewis JA, Meyer DE. Mind the Hype: A Critical Evaluation and Prescriptive Agenda for Research on Mindfulness and Meditation. Perspect Psychol Sci. 2018 Jan;13(1):36-61. doi: 10.1177/1745691617709589. Epub 2017 Oct 10. PMID 29016274
- [Background] Weinberger DR, Radulescu E. Structural Magnetic Resonance Imaging All Over Again. JAMA Psychiatry. 2021 Jan 1;78(1):11-12. doi: 10.1001/jamapsychiatry.2020.1941. No abstract available. PMID 32697315
- [Background] Boubela RN, Kalcher K, Huf W, Seidel EM, Derntl B, Pezawas L, Nasel C, Moser E. fMRI measurements of amygdala activation are confounded by stimulus correlated signal fluctuation in nearby veins draining distant brain regions. Sci Rep. 2015 May 21;5:10499. doi: 10.1038/srep10499. PMID 25994551
- [Background] Turner R. How much cortex can a vein drain? Downstream dilution of activation-related cerebral blood oxygenation changes. Neuroimage. 2002 Aug;16(4):1062-7. doi: 10.1006/nimg.2002.1082. PMID 12202093
- [Background] Greene DJ, Black KJ, Schlaggar BL. Considerations for MRI study design and implementation in pediatric and clinical populations. Dev Cogn Neurosci. 2016 Apr;18:101-112. doi: 10.1016/j.dcn.2015.12.005. Epub 2015 Dec 17. PMID 26754461
- [Background] Kjaer TW, Bertelsen C, Piccini P, Brooks D, Alving J, Lou HC. Increased dopamine tone during meditation-induced change of consciousness. Brain Res Cogn Brain Res. 2002 Apr;13(2):255-9. doi: 10.1016/s0926-6410(01)00106-9. PMID 11958969
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Tang YY, Ma Y, Wang J, Fan Y, Feng S, Lu Q, Yu Q, Sui D, Rothbart MK, Fan M, Posner MI. Short-term meditation training improves attention and self-regulation. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17152-6. doi: 10.1073/pnas.0707678104. Epub 2007 Oct 11. PMID 17940025
- [Background] Carlson LE, Brown KW. Validation of the Mindful Attention Awareness Scale in a cancer population. J Psychosom Res. 2005 Jan;58(1):29-33. doi: 10.1016/j.jpsychores.2004.04.366. PMID 15771867
- [Background] Lazar SW, Kerr CE, Wasserman RH, Gray JR, Greve DN, Treadway MT, McGarvey M, Quinn BT, Dusek JA, Benson H, Rauch SL, Moore CI, Fischl B. Meditation experience is associated with increased cortical thickness. Neuroreport. 2005 Nov 28;16(17):1893-7. doi: 10.1097/01.wnr.0000186598.66243.19. PMID 16272874